CLINICAL TRIAL: NCT05895812
Title: A Non-Random, Open-label, Parallel-group Study to Assess the Pharmacokinetics of JT001 in Subjects With Mild and Moderate Renal Impairment Compared to Subjects With Normal Renal Function
Brief Title: A Study in Subjects With Renal Impairment Compared to Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JT001-008-I
Record Dates: First submitted 2023-05-15; First posted 2023-06-09 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-05

CONDITIONS: Subjects With Renal Impairment; Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Mild Renal Impairment
  Interventions: Drug: Deuremidevir Hydrobromide Tablets
- Arm 2 (Experimental): Moderate Renal Impairment
  Interventions: Drug: Deuremidevir Hydrobromide Tablets
- Arm 3 (Experimental): Healthy subjects
  Interventions: Drug: Deuremidevir Hydrobromide Tablets

INTERVENTIONS:
Drug: Deuremidevir Hydrobromide Tablets — JT001 single dose, 0.3g

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of a single dose of JT001 in adult subjects with mild and moderate renal impairment compared to healthy mean-matched subjects.The results of this study will guide the clinical recommendation regarding whether or not a dose adjustment may be needed when treating patients with renal impairment.

DETAILED DESCRIPTION:
This study will compare the pharmacokinetics of JT001 in patients with normal, mild or moderate renal impairment.There are 3 periods in the study including screening(D-28~D-1 prior to investigation product administration) 、treatment and assessment (D1~D4 domiciled in study center) and telephone follow-up(D7).

Twenty-four males and female volunteers between 18-65 years of age with BMI between 19- 28 kg/m2 will be divided into 3 groups of 8 subjects each based on renal function as defined (8 normal, 8 mild impairment, 8 moderate impairment).Participants in the renal impairment groups will be staged by their respective degree of renal function (mild or moderate) according to the estimated glomerular filtration rate (eGFR) determined at the screening visit. In order to exclude other factors that may affect the nature of PK, each renal impairment participant must be matched to a healthy control participant with respect to gender、age (±10 years) and body weight (±10kg).The subjects received a single dose of JT001 and collected blood and urine samples before and after administration for pharmacokinetic analysis.

After enrollment,subjects will be confined to the study unit during the entire 4 day study period.On day 1, after a fast of at least 10 hours, each patient will receive a single oral dose 0.3g of JT001. Blood and urine samples will be collected at times sufficient to adequately define the pharmacokinetics of JT001 active metabolite(116N-1) in the three study groups. Subjects will be monitored regarding adverse effects throughout study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form before the experiment and have a thorough understanding of the content, process, and potential adverse reactions of the experiment;
2. 18 years old ≤ age ≤ 65 years old, regardless of gender;
3. Body mass index (BMI) within the range of 19 kg/m2 to 28 kg/m2 (including both end values);
4. Subjects with renal insufficiency:

   The estimated glomerular filtration rate (eGFR, calculated using the CKD-EPI formula (refer to Attachment 3)) must meet the following criteria:

   Subjects with mild renal insufficiency (CKD2 stage): 60-89 mL/min/1.73m2 (including both end values) Subjects with moderate renal insufficiency (CKD3 phase): 30-59 mL/min/1.73m2 (including both end values)

   Healthy subjects:

   estimated Glomerular filtration rate (eGFR, calculated using the CKD-EPI (refer to Appendix 3) formula) ≥ 90 mL/min/1.73m2;
5. Subjects with renal insufficiency: The renal function status is stable, and the eGFR results of the two tests before administration (with an interval of at least 3 days between the two tests) must be within the same CKD stage;

Exclusion Criteria:

Subjects with renal insufficiency who meet any of the following criteria will not be eligible for admission to this study:

1. had a kidney transplant before;
2. Kidney dialysis is required during the study period;
3. Urinary incontinence or anuria;
4. Individuals who are allergic to research drugs or excipients;
5. Having clinically significant heart disease within 12 months prior to the start of treatment, including but not limited to: congestive heart failure, symptomatic coronary artery disease, myocardial infarction, QTcF ≥ 470 ms (female) or 450 ms (male), etc;
6. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 × ULN), or screening for clinically significant bleeding symptoms or clear bleeding tendencies within the first 3 months, such as gastrointestinal bleeding, hemorrhagic gastric ulcers, or undergoing thrombolytic and anticoagulant treatment;
7. Patients with hypertension, diabetes, hyperlipidemia and other basic diseases, who cannot be well controlled after drug treatment (including systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg);
8. Used 14 days before taking the study drug, or needed to be used during the test, any drug that affects the secretion of gastric acid, including but not limited to cimetidine, ranitidine, famotidine, rosatidine, nizatidine, omeprazole, lansoprazole, pirenzepine, rabeprazole, pantoprazole, aluminum hydroxide, etc; Or any Chinese medicine or traditional Chinese patent medicines and simple preparations needs to be used after signing the informed consent form to the end of PK blood collection;

Healthy subjects who meet any of the following criteria are not eligible to participate in this study:

1. Those who have definite diseases such as central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders, etc. and need medical intervention or other diseases that are not suitable for clinical trials (such as psychiatric history, etc.);
2. Those who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health products within the first 2 weeks of screening;
3. Those who are screened positive for urinary drug abuse, or have a history of drug abuse within the past five years or have used drugs in the past three months before the trial;
4. Positive individuals for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (Anti HCV), treponema pallidum antibody, and acquired immunodeficiency syndrome (HIV) antibody;
5. Abnormal chest X-ray (posterior anterior position) results with clinical significance;
6. B-ultrasound examination shows moderate to severe fatty liver disease;
7. When screening or baseline alanine transaminase (ALT) or aspartate transaminase (AST) exceeded the upper limit of normal value (ULN);
8. During screening or baseline electrocardiogram abnormalities, QTcF (corrected for heart rate) in a single examination for males>450 ms, females>470 ms, and/or other clinically significant abnormalities;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact on the Cmax of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  maximum observed plasma concentration
Evaluate the impact on the AUC0-t of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  area under the plasma concentration time curve from time zero to the last measurable concentration
Evaluate the impact on the AUC0-inf of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  area under the plasma concentration-time curve from time zero to infinity
Tmax of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  Evaluate the impact on the Tmax of the main metabolite 116-N1 of JT001;
t1/2 of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  Evaluate the impact on the t1/2 of the main metabolite 116-N1 of JT001;
CL/F of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  Evaluate the impact on the CL/F of the main metabolite 116-N1 of JT001;
Vz/F of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  Evaluate the impact on the Vz/F of the main metabolite 116-N1 of JT001;
Ae of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  Evaluate the impact on the Ae of the main metabolite 116-N1 of JT001;
CLr of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  Evaluate the impact on the CLr of the main metabolite 116-N1 of JT001;
Ae% of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  Evaluate the impact on the Ae% of the main metabolite 116-N1 of JT001;

SECONDARY OUTCOMES:
The incidence and severity of adverse events (TEAEs) of serious adverse events (SAE) occurred during the treatment were observed. | From Day 1(first dose) to Day7
  The incidence and severity of adverse events (TEAEs) of serious adverse events (SAE) occurred during the treatment were observed.
The incidence and severity of adverse events (TEAEs) of clinical symptoms occurred during the treatment were observed. | From Day 1(first dose) to Day7
  The incidence and severity of adverse events (TEAEs) of clinical symptoms occurred during the treatment were observed.
The incidence and severity of adverse events (TEAEs) of vital signs occurred during the treatment were observed. | From Day 1(first dose) to Day7
  The incidence and severity of adverse events (TEAEs) of vital signs occurred during the treatment were observed.
The incidence and severity of adverse events (TEAEs) of physical examination occurred during the treatment were observed. | From Day 1(first dose) to Day7
  The incidence and severity of adverse events (TEAEs) of physical examination occurred during the treatment were observed.
The incidence and severity of adverse events (TEAEs) of laboratory examination occurred during the treatment were observed. | From Day 1(first dose) to Day7
  The incidence and severity of adverse events (TEAEs) of laboratory examination occurred during the treatment were observed.
The incidence and severity of adverse events (TEAEs) of abnormal electrocardiogram (ECG) occurred during the treatment were observed. | From Day 1(first dose) to Day7
  The incidence and severity of adverse events (TEAEs) of abnormal electrocardiogram (ECG) occurred during the treatment were observed.

CONTACTS AND LOCATIONS:
Overall Officials: Huiyu Lan, Project Director, Study Director — Shanghai Vinnerna Biosciences Co., Ltd.
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided